CLINICAL TRIAL: NCT02684318
Title: Phase Ib/II Study to Evaluate the Efficacy and Tolerability of PM01183 in Combination With Olaparib in Patients With Advanced Solid Tumors
Brief Title: Study to Evaluate PM01183 in Combination With Olaparib in Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poveda, Andrés, M.D. (Individual)
Collaborators: AstraZeneca (Industry); PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POLA/ACOG1401
Record Dates: First submitted 2016-02-02; First posted 2016-02-18 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Advanced Cancer; Ovarian Cancer; Endometrial Cancer; Breast Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Breast Neoplasms | interventions — PM 01183; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Dose Level 1 (Experimental): PM01183 + olaparib PM01183: 1 mg/m² IV olaparib 100 mg BID
  Interventions: Drug: PM01183 + olaparib
- Dose Level 2 (Experimental): PM01183 + olaparib PM01183: 1 mg/m² IV olaparib 150 mg BID
  Interventions: Drug: PM01183 + olaparib
- Dose Level 3 (Experimental): PM01183 + olaparib PM01183: 1.5 mg/m² IV olaparib 200 mg BID
  Interventions: Drug: PM01183 + olaparib
- Dose Level 4 (Experimental): PM01183 + olaparib PM01183: 1.5 mg/m² IV olaparib 250 mg BID
  Interventions: Drug: PM01183 + olaparib
- Dose Level 5 (Experimental): PM01183 + olaparib PM01183: 2 mg/m² IV olaparib 250 mg BID
  Interventions: Drug: PM01183 + olaparib
- Dose Level 6 (Experimental): PM01183 + olaparib PM01183: 2 mg/m² IV olaparib 300 mg BID
  Interventions: Drug: PM01183 + olaparib
- Dose Level 7 (Experimental): PM01183 + olaparib PM01183 3 mg/m² IV olaparib 300 mg BID
  Interventions: Drug: PM01183 + olaparib

INTERVENTIONS:
Drug: PM01183 + olaparib
  Other Names: Lynparza; Lurbinectedin

SUMMARY:
Phase Ib/II study to evaluate the efficacy and tolerability of PM01183 in combination with olaparib in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The study will be split into 2 parts: an open label Phase I dose escalation part followed by a non-randomized Phase II part, as an expansion study, in patients with selected tumors at the recommended doses and schedule determined in the phase I.

Phase I: A dose escalation study will be performed in patients with advanced or metastatic solid tumors without established standard therapeutic alternatives.

Phase II: An expansion dose study selecting patients with potential tumors with possibly sensitivity to PARP inhibitors according to histology, including triple negative breast cancer, high grade serous platinum-resistant ovarian and endometrial cancer patients, or patients with molecular features such as endometrial cancer with PTEN loss, breast or ovarian cancer with PTEN loss, known BRCA1/2 germline, somatic mutation or somatic methylation.

OBJECTIVES:

Primary objectives:

Phase Ib: To establish the safety [dose limiting toxicity (DLT), maximum tolerated dose (MTD) and recommended Phase II doses (RP2D)], of orally administered olaparib in combination with PM01183 in patients with advanced or metastatic solid tumors without established standard therapeutic alternatives.

Phase II: To assess the efficacy in terms of Tumor response rate according to RECIST v1.1 criteria of PM01183 in combination with olaparib in the selected populations.

Secondary objectives

Phase Ib:

To explore the pharmacokinetics of PM01183 and olaparib when administered in combination. To determine the effects of the study treatment on the level of PARP activity and

DNA damage in:

* Peripheral blood mononuclear cells (PBMC).
* Circulating tumor cells (CTC).
* Tumor biopsy samples. To evaluate the preliminary antitumor activity (overall response rate) by RECIST of the combination in the exposed population.

Phase II:

Progression free survival. Overall Survival. Toxicity profile of the combination in patients enrolled in the study. To explore the possible correlation between the expression of certain biomarkers and the efficacy of this therapeutic approach.

STATISTICAL PROCEDURES

- Sample size. Justification

Phase I:

Between 18-48 patients are expected to participate in the Phase Ib part of the study. The number of patients may vary depending upon the tolerability of the combination and the number of dose levels required to identify the MTD.

Phase II:

A total accrual up to 73 subjects would be required, according to an MinMax two-stages Simon design. With an α-error 0.05 and a power 90%, RR with a poor scenario according previous one would be 24%, and in a favourable scenario RR would reach 40%.

Progression-free survival according to previous reported is 3.5 months and the objective for the study is 6.5 months (n=56). According to this objective, the maximum sample size is 73 patients, and first sample size is 61 patients (upper limit for first stage rejection: 18).

Two stages are established:

1. In the first step 61 evaluable patients will be included in the study. If 18 or fewer responses are observed, the study will be stopped due to an inadequate response rate.

   Efficacy data for the patients included at this first step will be reviewed by an independent assessment committee (IAC).
2. If 19 or more responses are observed recruitment will continue until the group has 73 evaluable patients. If 23 or fewer responses are detected among these 73 patients, it will be concluded that the regimen is not sufficiently active to warrant further testing. If 24 or more responses are observed it will be concluded that the regimen is sufficiently active to warrant further testing in posterior Phase III.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age, no upper age limit.
* Written informed consent obtained prior to any study specific procedures or assessments.
* Histologically confirmed diagnosis of cancer:

  1. Phase I: patients with advanced or metastatic solid tumors without established standard therapeutic alternatives.
  2. Phase II: platinum-resistant ovarian cancer patients (epithelial non-mucinous), triple negative breast cancer and endometrial cancer (any grade).
* For patients included in the phase II part of the study, evidence of measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1 is required.

  1. At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements, OR
  2. At least one lesion (measurable and/or non-measurable) that can be accurately assessed by (CT/MRI/plain x-ray) at baseline and follow up visits.
* Patients included in the phase II part of the study must have received at least one line of standard therapy for locally advanced or metastatic disease, and developed progression disease afterwards.
* ECOG score < 2.
* Life expectancy of ≥ 3 months.
* Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

  1. Haemoglobin ≥ 10.0 g/dL and no blood transfusions in the 28 days prior to entry/randomisation (choose whichever is most applicable to the study).
  2. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L

  i. No features suggestive of myelodisplastic syndrome (MSD)/ Acute myeloid leukaemia (AML) on peripheral blood smear c. White blood cells (WBC) > 3x109/L d. Platelet count ≥ 100 x 109/L e. Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) f. AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional ULN unless liver metastases are present in which case it must be ≤ 5x ULN g. Albumin ≥ 3.0 g/dl h. Serum creatinine ≤ 1.5 x institutional ULN i. Creatinine clearance ≥ 30 ml/min.
* Patients should sign an informed consent form before inclusion in the study that specifies that the clinical trial treatment entails consent for the analysis of biological samples of tumor and blood.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Evidence of non-childbearing status for women of childbearing potential (WOCBP)*.

WOCBP should only be included after a confirmed menstrual period and a negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1.. The inclusion of WOCBP requires use of a highly effective contraceptive measure (Appendix H).

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

* Involvement in the planning and/or conduct of the study.
* Previous enrolment or randomization in the present study.
* Simultaneous participation in any other study involving an investigational medicinal product, or having participated in a study less than 28 days prior to the start of study treatment.
* For patients included in the phase I of the study, previous treatment with olaparib or PM01183. For patients included in the phase II of the study, any previous treatment with a PARP inhibitor, including olaparib, or PM01183.
* Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 2 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment with study drug.
* Olaparib and PM01183 are metabolized mainly by CYP3A4. Therefore, concomitant use of known strong CYP3A4 inhibitors such as ketokonazole, itraconazole, telithromycin and clarithromycin are forbidden. Concomitant use of known CYP3A4 strong inducers. (See Appendix K for a list of CYP inducers, inhibitors and substrates).
* Persistent toxicities (≥ CTCAE grade 2) with the exception of alopecia, caused by previous cancer therapy.
* Resting ECG with QTc > 470msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
* Patients with myelodysplastic syndrome/acute myeloid leukaemia.
* Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 28 days prior to treatment.
* Major surgery within 14 days of starting study treatment and patients must have recovered from any effects of any major surgery. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, unstable spinal cord compression (untreated and unstable for at least 28 days prior to study entry), superior vena cava syndrome, extensive bilateral lung disease on HRCT scan or any psychiatric disorder that prohibits obtaining informed consent.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Breast feeding women.
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV) and are receiving antiviral therapy.
* Patients with known active hepatic disease (i.e., Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids.
* Patients who present any contraindication or suspected allergy to the products (or any of the excipients) under investigation in the study.
* Patients with uncontrolled seizures.
* For patients included at the phase II part of the study: patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated insitu cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | 1 year
  To establish the Dose Limiting Toxicity in the dose escaltion study phase I
Maximum tolerated dose | 1 year
  To establish the Maximum tolerated dose in the dose escaltion study phase I
Efficacy in terms of Tumor Response Rate according to RECIST 1.1 criteria. | 3 years
  to assess the efficacy in terms of Tumor response rate according to RECIST 1.1 criteria of PM01183 in combination with olaparib in the selected populations

SECONDARY OUTCOMES:
Pharmacodynamic evaluation to assess the increasing activity in DNA damage | 1 year
  Pharmacodynamic evaluation to assess the increasing activity in DNA damage of the combination of PM01183+Olaparib ((double strand break).
Overall response rate | 3 years
  To evaluate the preliminary antitumor activity (overall response rate) by RECIST of the combination in the exposed population.
Progression free survival. | 3 years
  The time from inclusion until objective tumor progression or death from any cause.
Biomarker analysis | 3 years
  To explore the possible correlation between the expression of certain biomarkers and the efficacy of this therapeutic approach.
To demonstrate the predictive capacity and prognostic impact of some of the biomarkers under study. | 3 years
  * In peripheral blood:
    * Germline DNA: confirmation of HRD tumor findings if necessary.
    * PBMC: γH2AX (0 and X h after olaparib: to be defined after phase I findings) in the first cycle.
  * In archival tumor:
    * HRD panel by NGS.
    * BRCA1 methylation.
    * PTEN deficiency by IHC and/or FISH.
    * PTEN, BRCA1/2 mutation.
    * Tissue array to analyse other biomarkers by IHC (BRCA1 and other HRD genes).
  * In biopsy before study entry (limited to 15 patients):
    * IHC (RAD-51, PARP, γH2AX, PTEN, BRCA1).
    * PTEN, BRCA1/2 mutation.
    * Tissue array to analyze other immunohistochemical biomarkers (BRCA1 and other HRD genes).
  * In biopsy before study entry (limited to 15 patients):
    * IHC (RAD-51, PARP, γH2AX, PTEN, BRCA1).

CONTACTS AND LOCATIONS:
Overall Officials: Andres Poveda, MD, Principal Investigator — Fundación Instituto Valenciano de Oncología
Locations (6):
- Spain (6):
  - Hospital Reina Sofía, Córdoba, Andalusia
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Ramón y Cajal, Madrid
  - Hospital La Paz, Madrid
  - Fundación Instituto Valenciano de Oncología, Valencia

IPD SHARING:
Plan to Share IPD: No